CLINICAL TRIAL: NCT00002152
Title: Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of WF 10 IV Solution ( TCDO ) in the Management of Patients With Advanced HIV Disease
Brief Title: A Study of WF 10 IV Solution in Patients With Advanced HIV Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxo Chemie GmbH (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 222B; WF10-94-US-002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: WF10

SUMMARY:
The purpose of this study is to see if it is safe and effective to give WF 10 (TCDO) to patients with advanced HIV disease who cannot or will not take zidovudine, didanosine, zalcitabine, or stavudine. This study also examines how TCDO affects the levels of HIV in the body. TCDO is a solution delivered through a vein.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Approved drugs at a stabilized dose except those specifically excluded.
* Aerosolized pentamidine (300 mg) once a month for PCP prophylaxis.

Patients must have:

* HIV positivity.
* Absolute CD4 count < 200 cells/mm3.
* Intolerance to or refusal to take AZT, ddI, ddC, or d4T.
* No active opportunistic infection requiring ongoing therapy.
* Life expectancy at least 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Neoplasm other than basal cell carcinoma of the skin.
* Clinically significant cardiac disease.
* Anemia.

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapy.
* Corticosteroids.

Patients with the following prior conditions are excluded:

History of myocardial infarction or arrhythmias.

Prior Medication:

Excluded within 2 weeks prior to study entry:

* Any antiretroviral agent.
* Interferon.
* Systemic therapy with biologic response modifiers, corticosteroids, cytotoxic chemotherapy, or neutropenic or nephrotoxic drugs.

Excluded within 30 days prior to study entry:

* Investigational drugs.

Prior Treatment:

Excluded within 2 weeks prior to study entry:

* Radiation therapy. Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (1):
- Nashville Health Management Foundation / Vanderbilt Univ, Nashville, Tennessee, United States

REFERENCES:
- [Background] Kahn JO, McGrath MS, Ching OM, Kuhne FW. A single center, phase 2 study evaluating the effects of WF10. Int Conf AIDS. 1998;12:349 (abstract no 22423)
- [Background] Busch HW, Christensen S, Reichelt D, Jahn S, Zidek W. Treatment of HIV-infected patients with advanced symptomatic disease with WF10 solution (TCDO). Int Conf AIDS. 1994 Aug 7-12;10(1):204 (abstract no PB0245)
- [Background] Raffanti SP, Schaffner W, Federspiel CF, Blackwell RB, Ching OA, Kuhne FW. Randomized, double-blind, placebo-controlled trial of the immune modulator WF10 in patients with advanced AIDS. Infection. 1998 Jul-Aug;26(4):202-7. doi: 10.1007/BF02962364. PMID 9717676